CLINICAL TRIAL: NCT03332758
Title: Inflammasomes in Cell Death in Macular Hole, Epiretinal Membrane, and Rhegmatogenous Retinal Detachment
Brief Title: Inflammasomes in Cell Death in FTMH, ERM, and RRD
Status: Completed | Type: Observational
Sponsor: Allen C. Ho, MD (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Sponsor-Investigator, Allen C. Ho, MD, Principal Investigator, Wills Eye
Organization: Wills Eye (Other)
Other Study IDs: 17-660E
Record Dates: First submitted 2017-10-13; First posted 2017-11-06 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Retinal Detachment; Full Thickness Macular Hole; Epiretinal Membrane
Keywords: retinal detachment; inflammasome; macular hole
MeSH Terms: conditions — Retinal Detachment; Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vitreous fluid and subretinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- RD treated with vitrectomy: Vitreous fluid from retinal detachment treated with pars plana vitrectomy
  Interventions: Procedure: Pars plana vitrectomy
- RD treated with external drainage: Subretinal fluid from retinal detachment treated with external drainage.
  Interventions: Procedure: External drainage
- Macular holes treated with vitrectomy: Vitreous fluid from patients treated for macular hole
  Interventions: Procedure: Pars plana vitrectomy
- ERM treated with vitrectomy: Vitreous fluid from patients treated for epiretinal membrane
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — Standard of care treatment for retinal detachment, macular hole, or epiretinal membrane.
  Groups: ERM treated with vitrectomy; Macular holes treated with vitrectomy; RD treated with vitrectomy
Procedure: External drainage — Standard of care treatment for retinal detachment.
  Groups: RD treated with external drainage

SUMMARY:
Prospective study evaluating the role of inflammasomes in cell death in retinal detachment, full thickness macular hole, and epiretinal membrane. The investigators are collecting vitreous and subretinal fluid samples from patients with these conditions and evaluating activity of the inflammasome pathway with established assays.

DETAILED DESCRIPTION:
Photoreceptor cell death is the main cause of vision loss in many retinal disorders, including retinal detachment (RD). While apoptosis is the most studied form of cell death, the investigators believe patients with RDs may have photoreceptor cell death from a distinct pathway of programmed cell death called pyroptosis which also involves an inflammatory response. Pyroptosis is distinct from apoptosis in that it requires the activation of a protein oligomer complex called an inflammasome. The inflammasome is a pro-inflammatory complex composed of apoptosis-associated speck-like protein containing a CARD (ASC), nucleotide-binding oligomerization domain-containing protein (NOD)-like receptor (NLR) family or pyrin and HIN domain (PYHIN) family, and caspase-11. Activation of the inflammasome complex leads to activation of capspase 1 proteolytic activity to cleave and synthesize IL-1β and IL-18. As such the investigators believe inflammasomes and its activated products may play a strong role in the inflammatory and cell death pathway for photoreceptor cells in human retina. Studies using animal models of RD have already confirmed the presence of IL-1β activation2, however, the presence of IL-18 needs to be confirmed in human detached retinas. In a study performed on the detached retinas in mice, researchers were able to show activation of inflammasomes leading to photoreceptor cell death. While researchers are unable to determine the cellular source of the inflammasomes they were able to show that activation inflammasomes closely follows animal models. Currently there is no method to rescue photoreceptors cells from the mediated cell death pathway despite surgical intervention. Thus, current visual prognosis and prevention of further photoreceptor loss due to a RD is likely dependent on the time of surgical intervention before further detachment and further cell death can occur. As such, the purpose of this current study is to confirm the presence of inflammasome activation as well as the synthesis of its products, IL-1β and IL-18, in patients with rhegmatogenous retinal detachments. Both inflammasomes and its products IL-1β and IL-18 may be involved in cell pyroptosis, a programmed cell death distinct from apoptosis. Due to a lack of treatment for the rescue of photoreceptor cells from cell death after a retinal detachment, this study can provide novel strategies to inhibit cell death.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of the Wills Eye Hospital Retina service and Mid-Atlantic Retina offices.
2. Volunteer patients age 18 years and older.
3. Healthy enough to participate in the study.
4. Willing and able to consent to participation in the study.
5. Diagnosis of rhegmatogenous retinal detachment treated with external drainage of subretainl fluid, rhegmatogenous retinal detachment treated with pars plana vitrectomy, or full thickness macular hole treated with pars plana vitrectomy

Exclusion Criteria:

1. Presence of tractional retinal detachment
2. History of trauma
3. Presence of proliferative vitreoretinopathy
4. History of prior retinal detachment repair or any prior retina surgery or laser treatment e. Any preexisting retinal disease (including diabetic retinopathy, age related macular degeneration, retinal vein or artery occlusion, other retinal vascular disease, inherited retinal degeneration, uveitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with retinal detachment, macular hole, or epiretinal membrane.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Presence of inflammasomes and their active products | Day of surgery
  Presence of inflammasomes and their active products in patients with retinal detachment treated with vitrectomy or external drainage, macular holes treated with vitrectomy, and epiretinal membranes treated with vitrectomy

SECONDARY OUTCOMES:
Difference in inflammasome levels among samples | Day of surgery
  Difference in inflammasome pathway activation between retinal detachment, macular hole, and epiretinal membrane samples

CONTACTS AND LOCATIONS:
Overall Officials: Allen C Ho, MD, Principal Investigator — MidAtlantic Retina
Locations (1):
- MidAtlantic Retina-Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
manuscript under development

REFERENCES:
- [Background] Murakami Y, Notomi S, Hisatomi T, Nakazawa T, Ishibashi T, Miller JW, Vavvas DG. Photoreceptor cell death and rescue in retinal detachment and degenerations. Prog Retin Eye Res. 2013 Nov;37:114-40. doi: 10.1016/j.preteyeres.2013.08.001. Epub 2013 Aug 28. PMID 23994436
- [Background] Kataoka K, Matsumoto H, Kaneko H, Notomi S, Takeuchi K, Sweigard JH, Atik A, Murakami Y, Connor KM, Terasaki H, Miller JW, Vavvas DG. Macrophage- and RIP3-dependent inflammasome activation exacerbates retinal detachment-induced photoreceptor cell death. Cell Death Dis. 2015 Apr 23;6(4):e1731. doi: 10.1038/cddis.2015.73. PMID 25906154